CLINICAL TRIAL: NCT04078529
Title: Efficacy of a Tailored Exercise Programme and Home Evaluation for Falls Prevention in Older People With a Visual Impairment
Brief Title: Falls Prevention for Visually Impaired Older People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Blind Veterans UK (Other)
Responsible Party: Principal Investigator, Catherine Wood, Physiotherapist, Health and Wellbeing Dept., Blind Veterans UK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FPIS0.1
Record Dates: First submitted 2019-08-30; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Accidental Fall; Visual Impairment; Fall
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Intervention Model Description: Single-blind randomised control trial
Who Masked: Participant
Masking Description: Participants will be unaware whether they are in the comparison or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group will complete a 5 day falls prevention training programme, followed by a 12 week home exercise programme, then a repeat 5 day training intervention.
  Interventions: Other: 5 day falls prevention training; Other: Home exercise programme; Other: Environmental Assessment
- Comparison group[ (Active Comparator): This group will complete the home exercise programme only.
  Interventions: Other: Home exercise programme; Other: Environmental Assessment

INTERVENTIONS:
Other: 5 day falls prevention training — Intensive training on balance, gait re-education, functional activities, backwards chaining and postural control, completed at 0 and 12 weeks.
  Arms: Intervention group
Other: Home exercise programme — A modified version of the Falls Management Exercise programme (FaME) provided in written or audio format and completed over 12 weeks.
Other: Environmental Assessment — Use of the Homefast assessment tool to reduce risk of falls at home.

SUMMARY:
This study aims to examine the effectiveness of an intensive five day falls prevention training programme with a home evaluation and a home exercise programme, compared with a home evaluation and exercise programme alone for reducing incidence of falls and fear of falling, and improving confidence in functional ability and objective balance.

DETAILED DESCRIPTION:
While previous research shows a clear link between visual impairment and increased risk and incidence of falls, as well as fear of falling, there is little research to investigate the effectiveness of falls prevention programmes for visually impaired populations. At the time of writing there were no studies identified that used this type of intensive training over a period of several days, rather most of the studies that exist have been conducted in community settings.

This study will aim to compare the effectiveness of a comprehensive exercise programme aimed at improving balance, walking technique, postural control and ability to complete functional tasks, with a home exercise programme with either written or audio instructions.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to mobilise with or without walking aids or hand-hold
* Participant has history of falls
* Any possible medical or pharmaceutical causes of falls have been investigated and excluded
* Participant has a diagnosed visual impairment
* Participant is aged 65 or over
* Participant's falls can not be attributed purely to their visual impairment
* Participant is a member of Blind Veterans UK
* Participant is physically able to take part in group and individual exercise sessions
* Participant is able to understand and follow verbal and/or written instructions

Exclusion Criteria:

* Participant is under 65 years of age
* Participant is medically unwell or has a medical condition for which exercise is contraindicated
* Participant is currently involved in other falls prevention programmes
* Participant is predominantly a wheelchair user
* Participant is unable to understand or follow instruction from staff in English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in Incidence of falls | Fortnightly reporting throughout the 12 week programme.
  Participant's self-reported incidence of falls or near misses
Change in Fear of falling | Completed at the time of consent to participate in the study and at week 0 and week 12 of the programme
  The participant's self-reported level of fear about their risk of having a fall as indicated by completion of the Falls Efficacy Scale (FES-I), which scores from a minimum of 1 to a maximum of 4 on each item with a high score indicating a worse outcome. The lowest total score possible is 16 and the highest total score possible is 64.
Change in Objective Balance | At 0 and 12 weeks in the programme
  Standing balance as measured by the 4-point balance test

SECONDARY OUTCOMES:
Risk of falls | Completed at the time of consent to participate in the study and at week 0 and 12 in the programme.
  The participant's likelihood of experiencing a fall as measured by the Falls Risk Assessment Tool (FRAT), which scores from a minimum of 0 to a maximum of 5, with a higher score indicating a worse outcome.
Confidence in functional ability | Completed at weeks 0 and 12 of the programme.
  Self-reported confidence in ability to perform activities of daily living as recorded using the Activities-specific Balance Confidence (ABC) scale, which scores from a minimum of 0 to a maximum of 10 on each of the 16 items. An average is then taken from the scores, with a higher average indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Wood, MSc PT, Principal Investigator — Blind Veterans UK
Locations (1):
- Blind Veterans UK, Llandudno, Conwy, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjerk M, Brovold T, Skelton DA, Bergland A. Associations between health-related quality of life, physical function and fear of falling in older fallers receiving home care. BMC Geriatr. 2018 Oct 22;18(1):253. doi: 10.1186/s12877-018-0945-6. PMID 30348098
- [Background] Huang ZG, Feng YH, Li YH, Lv CS. Systematic review and meta-analysis: Tai Chi for preventing falls in older adults. BMJ Open. 2017 Feb 6;7(2):e013661. doi: 10.1136/bmjopen-2016-013661. PMID 28167744
- [Background] Cuevas-Trisan R. Balance Problems and Fall Risks in the Elderly. Phys Med Rehabil Clin N Am. 2017 Nov;28(4):727-737. doi: 10.1016/j.pmr.2017.06.006. PMID 29031339
- [Background] Skelton DA, Bailey C, Howel D, Cattan M, Deary V, Coe D, de Jong LD, Gawler S, Gray J, Lampitt R, Wilkinson J, Adams N. Visually Impaired OLder people's Exercise programme for falls prevenTion (VIOLET): a feasibility study protocol. BMJ Open. 2016 Aug 2;6(8):e011996. doi: 10.1136/bmjopen-2016-011996. PMID 27486124
- [Background] Graham V, Napier-Dovorany K. Multifactoral measures of fall risk in the visually impaired population: A pilot study. J Bodyw Mov Ther. 2016 Jan;20(1):104-109. doi: 10.1016/j.jbmt.2015.06.012. Epub 2015 Jul 3. PMID 26891644
- [Background] Yeung PY, Chan W, Woo J. A community-based Falls Management Exercise Programme (FaME) improves balance, walking speed and reduced fear of falling. Prim Health Care Res Dev. 2015 Apr;16(2):138-46. doi: 10.1017/S1463423614000024. Epub 2014 Jan 30. PMID 24480023
- [Background] Martin JT, Wolf A, Moore JL, Rolenz E, DiNinno A, Reneker JC. The effectiveness of physical therapist-administered group-based exercise on fall prevention: a systematic review of randomized controlled trials. J Geriatr Phys Ther. 2013 Oct-Dec;36(4):182-93. doi: 10.1519/JPT.0b013e3182816045. PMID 23449007
- [Background] Tricco AC, Thomas SM, Veroniki AA, Hamid JS, Cogo E, Strifler L, Khan PA, Robson R, Sibley KM, MacDonald H, Riva JJ, Thavorn K, Wilson C, Holroyd-Leduc J, Kerr GD, Feldman F, Majumdar SR, Jaglal SB, Hui W, Straus SE. Comparisons of Interventions for Preventing Falls in Older Adults: A Systematic Review and Meta-analysis. JAMA. 2017 Nov 7;318(17):1687-1699. doi: 10.1001/jama.2017.15006. PMID 29114830
- [Background] Klein PJ, Baumgarden J, Schneider R. Qigong and Tai Chi as Therapeutic Exercise: Survey of Systematic Reviews and Meta-Analyses Addressing Physical Health Conditions. Altern Ther Health Med. 2019 Sep;25(5):48-53. PMID 31221939
- [Result] Adams N, Skelton DA, Howel D, Bailey C, Lampitt R, Fouweather T, Gray J, Coe D, Wilkinson J, Gawler S, de Jong LD, Waterman H, Deary V, Clarke M, Parry SW. Feasibility of trial procedures for a randomised controlled trial of a community based group exercise intervention for falls prevention for visually impaired older people: the VIOLET study. BMC Geriatr. 2018 Dec 12;18(1):307. doi: 10.1186/s12877-018-0998-6. PMID 30541483